CLINICAL TRIAL: NCT01448356
Title: Controlled Adverse Environment: A Pilot Study to Evaluate Tear Film Stability and Tear Evaporation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Eye Research Institute (Other)
Collaborators: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Andrea Petznick, PhD, Postdoctoral Research Fellow, Singapore Eye Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R857/52/2011; 2011/197/A (Other: Singhealth Centralised Institutional Review Board)
Record Dates: First submitted 2011-10-04; First posted 2011-10-07 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-11

CONDITIONS: Environmental Exposure
Keywords: Controlled adverse chamber; tear film stability; tear film evaporation; tear film break up time; humidity; temperature
MeSH Terms: interventions — Temperature; Humidity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- temperature and humidity (Experimental): The volunteer is exposed to a controlled environment with a chamber setting of:
  1. 25°C and 45% humidity;
  2. 25°C and 65% humidity;
  3. 30°C and 45% humidity;
  4. 30°C and 65% humidity
  Interventions: Procedure: temperature and humidity

INTERVENTIONS:
Procedure: temperature and humidity — The volunteer is exposed to a controlled environment with a chamber setting of:
  1. 25°C and 45% humidity;
  2. 25°C and 65% humidity;
  3. 30°C and 45% humidity;
  4. 30°C and 65% humidity
  After an adaptation period of at least 20 minutes, participants underwent measurements of tear evaporation and tear film break up time. After collection of data, the chamber settings were adjusted to the next condition.

SUMMARY:
Dry eye and ocular surface disease account for a lot of morbidity and socio-economic burden in Asia and the rest of the world. This is a small pilot study to evaluate tear function under different conditions of humidity and temperature. This data will be useful for designing future trials in ocular surface and dry eye. The data will likely be used to propose a larger national funded project involving clinical trials. This study involves collaboration between engineers, ocular surface clinicians as well as specialists from the defence science organisation. When successfully completed, the project will increase the capability of Singapore Eye Research Institute and Singapore National Eye Centre to support future industry and academic research in the ocular surface.

DETAILED DESCRIPTION:
Study Objectives and Purpose:

1. A primary purpose of the study is to evaluate fluorescein tear break up times in participants under different humidity/ temperature conditions.
2. The second aim is to assess the tear evaporation rates in a dynamic fashion over 20 seconds (based on a non-invasive ocular thermography method) after exposure to different humidity/temperature conditions.

Study Design: Prospective, non-comparative, clinical study

Rationale:

The ocular surface research team who is based at the dry eye service of the Singapore National Eye Center is experienced in the assessment of the ocular surface in patients and clinical trial participants. Collaborators from the DSO National laboratory already have experience in conducting human studies in a controlled environment in Singapore that has been proven to be safe and has passed necessary regulatory approval. In addition, recent technological advances have allowed collaborators from NTU and Singapore Polytechnic to perform non-invasive tear evaporimetry in a dynamic way between blinks. Together, this is a strong research team that can address the important question of the influence of temperature and humidity on the tear film stability.

Methods:

We intend to use 10 volunteer/patients to establish whether tear film stability or tear film function can be altered after exposure to different combinations of humidity and temperature. This involves the assessment of tear film break up time (TBUT) and tear evaporimetry, a non-invasive procedure (like an auto-refractor where the patient places the chin on the chin rest and forehead on the head rest when the measurement is taken) which involves taking serial images with an infra red sensitive video camera. This process is performed at a facility which is closely monitored and proven to be safe for other research participants.

Participants and target sample size: Ten participants will be recruited.

Workflow:

We assume that approximately 45 minutes are required for the chamber to achieve the required temperature and humidity, and about 15 to 20 minutes for participants to adjust to the first environmental setting. Thermography measurement will take 1 minute (20 sec in each eye, with adjustment of camera between eyes). The participants will undergo slit lamp examination where the fluorescein tear break up time will be assessed and digital color image of the break up pattern will be taken. These will require a further 5 minutes. This means 3 participants can have measurements done in approximately 20 minutes. Measurements of 3 participants in a single condition will therefore take up to 20 minutes.In a session that will last up to 3 hours and 20 minutes, the investigators can complete the condition list for 3 participants. Since the overall session is quite long, a toilet break is permitted after each temperature condition.

The investigators estimate that 3 sessions with a further 'dry run' for the photography (without participants) before the first session will be necessary.

Visit schedules:

Volunteers or patients from the Singapore National Eye Center will be informed of this study. Screening will be performed at the regular dry eye clinic at the Singapore National Eye Center. If eligible, the volunteer or patient will sign consent and undergo baseline examination. Subsequent to this, the examination will be performed at the controlled adverse environment at the DSO facility.

Assessment of ocular parameters is outlined below:

At Screening visit, the investigators perform:

* Informed consent
* Subject background
* Anterior segment findings
* Tear film break up time

At Evaluation visit, the investigators perform:

* Tear film break up time
* Photography/Video to document tear break up
* Tear evaporimetry

Duration of study: Four weeks.

ELIGIBILITY:
Inclusion Criteria:

* must have undergone screening examination

Exclusion Criteria:

* unable to go to the DSO laboratory or undergo any of the study procedures

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Petznick, PhD, Principal Investigator — Singapore Eye Research Institute
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Gonzalez-Garcia MJ, Gonzalez-Saiz A, de la Fuente B, Morilla-Grasa A, Mayo-Iscar A, San-Jose J, Feijo J, Stern ME, Calonge M. Exposure to a controlled adverse environment impairs the ocular surface of subjects with minimally symptomatic dry eye. Invest Ophthalmol Vis Sci. 2007 Sep;48(9):4026-32. doi: 10.1167/iovs.06-0817. PMID 17724183
- [Background] Wolkoff P. Ocular discomfort by environmental and personal risk factors altering the precorneal tear film. Toxicol Lett. 2010 Dec 15;199(3):203-12. doi: 10.1016/j.toxlet.2010.09.001. Epub 2010 Sep 15. PMID 20833234

RESULTS

PARTICIPANT FLOW:
Groups:
- Temperature and Humidity: All conditions were tested in a CAE chamber on the same day.
Period: Overall Study
Arm/Group | Temperature and Humidity
Started | 10
Completed | 10 (cross-over)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Temperature and Humidity
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 20.4 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Region of Enrollment [Number; unit: participants]
  Singapore | 10

OUTCOME MEASURES:

1. Primary Outcome: Tear Evaporation Rate
Description: The rate of tear evaporation is measured by the use of ocular thermography. For each subject,his/her ocular surface temperature will be recorded twice, one for each eye. The subject at first rests his/her chin on a chin rest, with his/her forehead lean against a metal frame (which is part of the chin rest). Then the recording starts lasting approximately 20seconds for each eye. While recording, the subject needs to look straight into the lens, but can blink naturally. After this, the recording data will be analyzed to derive the evaporation rate using a mathematical model.
Time Frame: 20 minutes after the required temperature and humidity in the chamber is achieved
Measure: Mean (95% Confidence Interval); unit: Watt/meter^2
Groups:
- Temperature and Humidity: Tear evaporation of overall surface
Arm/Group | Temperature and Humidity
Number analyzed (Participants) | 10
Watt/meter^2
  25°C and 45% humidity | 39.0 [33.0 to 45.0]
  25°C and 65% humidity | 44.8 [39.4 to 50.3]
  30°C and 45% humidity | 30.6 [25.9 to 35.4]
  30°C and 65% humidity | 26.7 [21.3 to 32.0]

2. Secondary Outcome: Tear Film Break up Time
Description: After instillation of fluorescein, the participant will then be asked to open the eyes, look ahead at the observer's forehead and not blink for as long as possible. The break up time is defined as the time between the lid opening and the first appearance of any dry spot on the cornea. The participant will be requested to close his eyes for few seconds and the procedure will be repeated for the left eye.
Time Frame: 20 minutes after the required temperature and humidity in the chamber is achieved
Measure: Mean (95% Confidence Interval); unit: seconds
Groups:
- Temperature and Humidity: average of three measurements
Arm/Group | Temperature and Humidity
Number analyzed (Participants) | 10
seconds
  25°C and 45% humidity | 5.9 [4.0 to 7.7]
  25°C and 65% humidity | 4.4 [3.1 to 5.7]
  30°C and 45% humidity | 5.0 [3.2 to 6.9]
  30°C and 65% humidity | 4.6 [3.0 to 6.2]

ADVERSE EVENTS:
Arm/Group | Temperature and Humidity
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes